CLINICAL TRIAL: NCT06662214
Title: Nutrient Profile and Muscle Protein Synthesis in Response to Corn Bread Made From Refined Versus Whole Grain Maize Flour
Acronym: PRO-CORN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2224550
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Effect of Food
Keywords: muscle protein synthesis; post-prandial nutrient and hormonal profile; farming practices

STUDY DESIGN:
Intervention Model Description: Participants will consume a meal corn bread plus mung bean stew, which type (refined vs. whole grain) consumed will be randomized where neither the participant nor investigator will know which meal is being consumed. Each participant will repeat the protocol two times.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A randomized double-blind crossover design with neither the subjects nor the investigators knowing who is on which food. The interventions will be coded using a blinded alphabetical letter code (A, B). A delegate researcher (independent party not further involved in the study) will randomize all interventions using a computer-generated randomization list. The delegate will hand in the code-breaker to the principal investigator in a sealed envelope. The envelope will be stored in a locked filing cabinet in the principal investigator's office, which will also be locked when unoccupied. The envelope will be opened by the principal investigator after completing the analysis of blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Refined maize flour (Experimental): This arm will be given a meal of corn bread made from refined maize flour and a portion of the mung bean stew meat together with 250mL of water
  Interventions: Other: Refined maize flour
- Whole grain flour (Experimental): This arm will be given a meal of corn bread made from whole grain maize flour and a portion of the mung bean stew meat together with 250mL of water
  Interventions: Other: Whole grain flour

INTERVENTIONS:
Other: Refined maize flour — Meal made form refined maize flour
  Arms: Refined maize flour
Other: Whole grain flour — Meal made form whole grain maize flour
  Arms: Whole grain flour

SUMMARY:
The purpose of the study is to quantify and compare the serum nutrient and hormonal profile, and muscle protein synthesis rates, in response to consuming isonitrogenous amounts of a traditional East African meal, mung bean stew with a traditional African corn bread made from two different kinds of maize (whole corn flour or refined).

Specific aim 1: Describe the post-prandial nutrient and hormonal profile in serum in the 3 hours following consumption of a portion of mung bean stew with traditional African corn bread made with either whole grain maize flour or refined maize flour.

Specific aim 2: Compare the ability a portion of mung bean stew and traditional African corn bread made with either whole grain maize flour or refined maize flour to activate mTORC1-specific and whole muscle protein synthesis in an in vitro model of muscle.

DETAILED DESCRIPTION:
Indicators of longevity in humans include skeletal muscle mass and strength. Muscle mass is determined by the balance between myofibrillar protein synthesis and degradation, influenced by diet and physical activity. Muscle strength is closely tied to muscle mass, and activities like weight lifting until failure have been shown to increase muscle protein synthesis, enhancing muscle mass and strength over time. Protein intake is essential for maintaining a positive protein balance and promoting muscle growth. While animal proteins are generally more effective than plant proteins at promoting muscle protein synthesis, many cultures rely on staple plant-based foods, such as maize, rather than animal-based protein sources.

Maize (Zea mays) flour is a leading staple in African diets, where it is consumed in various forms, including porridges and breads like Ugali in East Africa or Fufu in West Africa. The nutritional profile of this corn bread varies greatly depending on whether it is made with refined or whole-grain maize flour. Whole-grain maize flour retains the bran, germ, and endosperm, providing higher fiber, vitamins, and minerals, while refined maize flour primarily contains the endosperm. Although refined maize is lower in fiber, it has a higher proportion of the leucine-rich zein, a major corn protein. These nutritional differences could significantly impact metabolism and overall health.

Given that approximately a fifth of the global population relies on corn meal as a dietary staple, understanding the impact of refined versus whole-grain maize flour on muscle protein synthesis and serum amino acid content could provide valuable insights for dietary guidelines and public health. This study aims to explore these effects, comparing the post-meal nutrient profile and muscle protein synthesis response to traditional African corn bread made with whole-grain versus refined maize flour.

The purpose of the study is to quantify and compare the serum nutrient and hormonal profile and muscle protein synthesis rates in response to consuming isonitrogenous servings of traditional African corn bread made from whole-grain or refined maize flour, paired with mung bean stew.

Specific aim 1: Describe the post-prandial nutrient and hormonal profile in serum in the 3 hours following consumption of a portion of mung bean stew with traditional African corn bread made with either whole grain maize flour or refined maize flour.

Specific aim 2: Compare the ability a portion of mung bean stew and traditional African corn bread made with either whole grain maize flour or refined maize flour to activate mTORC1-specific and whole muscle protein synthesis in an in vitro model of muscle.

Study participants will attend the CTSC Clinical Research Center on two separate occasions.

The two study visits will be scheduled over a 2-week period (i.e., once per week for 2 weeks) at the same time in the morning after an overnight fast of more than 12 hours. Participants will be asked to refrain from vigorous exercise, caffeine, nicotine, and alcohol for 24 hours before each visit. Female participants will schedule their visits within the first two weeks of their menstrual cycle to control for hormone fluctuations that may affect digestion and metabolism.

Upon arrival at the research center for the first test visit, each participant's height and weight will be measured. They will also complete a questionnaire covering their physical activity and dietary habits.

I. Baseline blood draw.

Participants will be seated in individual testing rooms equipped with reclining phlebotomy armchairs. A nurse will insert a 22G catheter into a forearm vein to collect an initial 5 mL baseline blood sample.

II. Test meal.

After baseline blood collection, participants will consume one of the two corn bread test meals. The meal consists of a serving of mung bean stew and an isonitrogenous amount of either whole-grain or refined maize flour-based corn bread:

The food will be weighed before cooking, and an eighth of a teaspoon of salt will be added to enhance palatability and participants will be asked to consume the meal within a 10-minute period, chewing thoroughly. Participants will also drink a 250 mL glass of water with the meal.

III. Postprandial blood draws.

After the test meal, participants will remain at the research site in their testing rooms for 3 hours, where they may bring books or electronic devices to occupy themselves. Five additional 5 mL blood samples will be collected at 30, 60, 90, 120, and 180 minutes post-meal, totaling 30 mL per visit, and 60 mL for participants completing the study.

Blood samples will be collected in 5 mL serum-separating tubes. Samples will clot before centrifugation at 1000 x g for 10 minutes. The serum will then be frozen and stored at -80°C. One milliliter from each serum sample will be used to determine nutrient and hormone concentrations. The remainder will be used for muscle protein synthesis and mTORC1 bioassay analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy active males and females (To be considered active, volunteers must meet the following American College of Sports Medicine's guideline for physical activity for healthy adults: performing at least 150 minutes per week of moderate-to-vigorous intensity physical activity.
* Age18-30 years
* Normal weight (BMI between 18 and 25 kg/m2

Exclusion Criteria:

* Health or dietary restrictions that would prevent consumption of the test foods
* Known food allergy to corn
* Anemia (low red blood cell count)
* Overweight or obesity (BMI > 25 kg/m2)
* Receiving any medication that may interfere with the study
* Metabolic or endocrine disorder that would affect the digestion, absorption, and/or physiological response to any of the nutrients ingested.
* Currently not meeting the ACSM physical activity recommendations (IPAQ score < 150 min/week of moderate-to-vigorous physical activity.
* Pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
post-prandial amino acid profile | [Time Frame: Baseline (0 hour) to 30, 60, 90, 120 and 180 minutes after consumed meal]
  Serum samples are extracted with 1mL of modified Folch extraction, followed by vacuum centrifugation for drying. Dried samples will be reconstituted with 100 μl of 75% ACN/water. The supernatant is then injected into Aligent UPLC-QqQ for analysis of targeted free amino acids, short peptides, and other metabolites.
post-prandial short peptide profile | [Time Frame: Baseline (0 hour) to 30, 60, 90, 120 and 180 minutes after consumed meal]
  Serum samples are extracted with 1mL of modified Folch extraction, followed by vacuum centrifugation for drying. Dried samples will be reconstituted with 100 μl of 75% ACN/water. The supernatant is then injected into Aligent UPLC-QqQ for analysis of targeted free amino acids, short peptides, and other metabolites.
Muscle protein synthesis | [Time Frame: Baseline (0 hour) to 30, 60, 90, 120 and 180 minutes after consumed meal]
  To measure muscle protein synthesis, stably transfected C2C12 muscle cells with a plasmid (pcDNA3 luciferase) will be used. C2C12Luc cells will be plated in 24-well plates and differentiated over 4 days. Differentiated C2C12 cells will be fasted by washing with PBS and then treating them with Test Media (20% DMEM) for 15 minutes. Fasted muscle cells will then be treated with Test Media containing 10% baseline or fed serum (from blood samples at 30, 60, 90,120 and 180 minutes after meal) for 3 hours. Cells will be collected in passive lysis buffer and firefly luciferase activity will be determined.
mTORC1 specific protein synthesis | [Time Frame: Baseline (0 hour) to 30, 60, 90, 120 and 180 minutes after consumed meal]
  To measure the ability of meal of chicken (conventional or regenerative) to activate mTORC1, stably transfected C2C12 muscle cells with a plasmid (pcDNA3-TOP luciferase) where the luciferase mRNA contains a 5'TOP. 5'TOP mRNA, which specifically regulated by mTORC1 activity, will be used. Differentiated C2C12TOPLuc muscle cells in 24-well plates will be stimulated using the baseline or fed serum (from blood samples at 30, 60, 90,120 and 180 minutes after meal). The degree of mTORC1 activation will be determined as the difference in slopes between the baseline and fed sera.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis CTSC Clinical Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No